CLINICAL TRIAL: NCT06426199
Title: Arthroscope-Guided Intra-Articular Injection of Chitosan-Hyaluronate Gel Mixture Versus Hyaluronic Acid in the Treatment of TMJ Internal Derangement: A Randomized Controlled Clinical Trial
Brief Title: Chitosan-Hyaluronate Gel Mixture Vs Hyaluronic for Internal Derangement
Acronym: TMJ
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Collaborators: Misr International University (Other); University of Nizwa (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12345asdfg
Record Dates: First submitted 2024-05-12; First posted 2024-05-23 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-01

CONDITIONS: TMJ Disc Disorder
Keywords: TMD; Hyaluronic acid; Chitosan; Arthroscopy; Intra Articular Injection; TMJ
MeSH Terms: interventions — Hyaluronic Acid

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intra-Articular Injection of Hyaluronic Acid (Active Comparator): Arthroscope-guided intra-articular injection of Hyaluronic Acid in patients with TMJ anterior disc displacement without reduction.
  Interventions: Drug: Hyaluronic Acid
- Intra-Articular Injection of chitosan-hyaluronate gel mixture (Active Comparator): Arthroscope-guided intra-articular injection of chitosan-hyaluronate gel mixture in patients with TMJ anterior disc displacement without reduction
  Interventions: Drug: Chitosan-Hyaluronate Gel Mixture

INTERVENTIONS:
Drug: Chitosan-Hyaluronate Gel Mixture — The operation will be under GA. TMJ arthroscopy will performed by the same TMJ arthroscopy surgeon. Lysis and lavage will be performed in the upper joint space in all cases based on the triangulation technique with an inferolateral approach. The arthroscopic procedure will include lysis of adhesions, lavage, manipulation, and debridement of the upper joint space. A 1.9-mm arthroscope with a video monitoring and recording system and a 2.2-mm protective cannula sheath will be used for TMJ arthroscopy. Ringer's lactate will be used as irrigation fluid. Both groups will receive the same arthroscopic treatments. The injection of 2 ml of Chitosan-Hyaluronate Gel Mixture into affected joints will be performed. Needles will be removed after the injection sites and covered its sites with gauze dressing.
  Arms: Intra-Articular Injection of chitosan-hyaluronate gel mixture
Drug: Hyaluronic Acid — The operation will be under GA. TMJ arthroscopy will performed by the same TMJ arthroscopy surgeon. Lysis and lavage will be performed in the upper joint space in all cases based on the triangulation technique with an inferolateral approach. The arthroscopic procedure will include lysis of adhesions, lavage, manipulation, and debridement of the upper joint space. A 1.9-mm arthroscope with a video monitoring and recording system and a 2.2-mm protective cannula sheath will be used for TMJ arthroscopy. Ringer's lactate will be used as irrigation fluid. Both groups will receive the same arthroscopic treatments. The injection of 2 ml of Hyaluronic acid into affected joints will be performed. Needles will be removed after the injection sites and covered its sites with gauze dressing.
  Arms: Intra-Articular Injection of Hyaluronic Acid

SUMMARY:
This study is designed to assess the impact of injecting sodium hyaluronic acid versus a chitosan-hyaluronate hybrid gel into the upper compartment of the temporomandibular joint (TMJ) as a treatment for anterior disc displacement without reduction. The study will include patients diagnosed with Stage III or IV TMJ internal derangement (anterior disc displacement without reduction), as classified by Wilkes, with diagnoses confirmed through clinical symptoms and MRI evaluations. Participants will be randomly divided into two groups, both undergoing TMJ arthroscopy. In the first group, 2 ml of chitosan-hyaluronic acid hybrid gel will be injected into the affected joints, whereas in the second group, 2 ml of hyaluronic acid (HA) will be administered. The study will compare and analyze outcomes in both groups, focusing on pain during TMJ function, clicking sounds, the extent of maximum mouth opening, and maximum lateral jaw movement.

DETAILED DESCRIPTION:
This study will be a prospective randomized controlled clinical study on a convenience sample of patients who will be selected from the Department of Oral and Maxillofacial Surgery, Faculty of Dental Medicine, Suez University. Patients selected are whom will be diagnosed with TMJ internal derangement (anterior disk displacement without reduction Stage III, Stage IV Wilkes classification) based on clinical symptoms and MRI evaluations. Inclusion criteria will be adults aged between 25 - 50 years old, sufficient clinical and magnetic resonance imaging (MRI) data that could be obtained before and after the treatment. The exclusion criteria will be hematological or neurological diseases, inflammation or connective tissue diseases, head and neck malignancies, history of treatment of TMJ disease or history of craniofacial surgery not related to internal derangement treatment, insufficient clinical and MRI data.

Participants will be selected based on established criteria. A total sample size of 20 (10 in each group) was calculated to detect an effect size of about 1.33-1.34, with a power (1-β error) of 0.8 (80%) using a two-sided hypothesis test, with a significance level (α error) 0.05 for data [13]. All patients will undergo a preoperative clinical evaluation including Pain level on forced mouth opening using visual analogue scale (VAS), assessment of mean lateral jaw movements, assessment of TMJ clicking, assessment of maximum mouth opening (MMO), deviation of mandibular midline during mouth opening and closure. All patients will do a Magnetic resonance imaging (MRI) to evaluate the disc displacement.All patients will undergo conservative treatment as the first line of treatment in all TMJID cases. All patients will be under general anesthesia.

For both groups, the operation will be under GA and The skin surface of the pre-auricular region will be disinfected with povidone iodine solution. For both groups, TMJ arthroscopy will performed by the same TMJ arthroscopy surgeon. Lysis and lavage will be performed in the upper joint space in all cases based on the triangulation technique with an inferolateral approach. The arthroscopic procedure will include lysis of adhesions, lavage, manipulation, and debridement of the upper joint space. A 1.9-mm arthroscope with a video monitoring and recording system and a 2.2-mm protective cannula sheath will be used for TMJ arthroscopy. Ringer's lactate will be used as irrigation fluid. Both groups will receive the same arthroscopic treatments. In the first group, the injection of 2 ml of chitosan-hyaluronic acid hybrid gel into affected joints, while 2 ml of HA will be injected in to affected joints in the second group. Needles will be removed after the injection sites and covered its sites with gauze dressing. Postoperative care and instructions:

1. Medications:

   Brufen* as a nonsteroidal anti-inflammatory drug (NSAIDs) relieving muscle pain and swelling. Myofen* as a muscle relaxant especially for people who grind or clench their teeth help to relax tight jaw muscles.
2. Application hot & cold packs:

   All patients will be instructed to apply an ice pack to the side of his face and temple area for about 10 minutes. Also, simple stretching exercises for his or her jaw should be done. Application a warm towel or pack to the side of his face for about 5 minutes five times daily for 4 days.
3. Soft diet:

Soft food such as yogurt, mashed potatoes, cheese, soup, fish, cooked fruits and vegetables, beans, and grains should be eaten. In addition, food should be cut into small pieces. Avoid hard and crunchy foods like hard rolls, raw carrots, thick and large foods that need your mouth to open wide to fit the foods. Also, chewy sticky foods (like caramels and taffy) avoided too for next 10 days.

ELIGIBILITY:
Inclusion Criteria:

1. Patients were diagnosed with TMJ internal derangement (anterior disk displacement without reduction Stage III, Stage IV Wilkes classification) based on clinical symptoms and MRI evaluations.
2. Age 25 - 50 years old.

Exclusion Criteria:

1. Hematological or neurological diseases.
2. Inflammation or connective tissue diseases.
3. Head and neck malignancies.
4. History of treatment of TMJ disease or history of craniofacial surgery not related to ID treatment.
5. Insufficient clinical and MRI data.

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-01-17 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Joint Pain | 3 months
  Self-pain and function of the jaw assessment, with Visual Analogue Scale (VAS), ranging from 0 to 10 scales. This scale will be used for self-evaluation of the patients, to evaluate pain level and jaw dysfunction and compared with preoperative degree. Patients will be asked about the pain severity & dysfunction according to the VAS.
lateral excursion | 3 months
  Maximum lateral excursion, the distance from midline of upper & lower jaw will be measured with a digital caliper in mm.
TMJ sounds | 3 months
  measured by asking the patients to open and closed his mouth several times and clicking was recorded as present (early clicking, late clicking) or absent.
Maximum mouth opening | 3 months
  Maximum mouth opening (MMO), between upper & lower incisors will be measured during maximum opening with a digital caliber in mm.

CONTACTS AND LOCATIONS:
Locations (1):
- Suez University, Suez, Egypt

IPD SHARING:
Plan to Share IPD: No